CLINICAL TRIAL: NCT02172443
Title: Comparison of 18 mcg of Tiotropium Inhalation Capsules and Atrovent Metered Dose Inhaler (2 Puffs of 20 mcg) in a Double Blind, Double Dummy, Efficacy and Safety Study in Adults With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Comparison of Tiotropium Inhalation Capsules and Atrovent Metered Dose Inhaler (MDI) in a Efficacy and Safety Study in Adults With Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 205.232
Record Dates: First submitted 2014-06-20; First posted 2014-06-24 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Ipratropium

ARMS (2):
- tiotropium inhalation capsules (Experimental)
  Interventions: Drug: tiotropium inhalation powder capsules; Drug: placebo to tiotropium inhalation capsules
- Atrovent MDI (Active Comparator)
  Interventions: Drug: Atrovent; Drug: placebo to Atrovent

INTERVENTIONS:
Drug: tiotropium inhalation powder capsules
  Arms: tiotropium inhalation capsules
Drug: Atrovent
  Arms: Atrovent MDI
Drug: placebo to Atrovent
  Arms: Atrovent MDI
Drug: placebo to tiotropium inhalation capsules
  Arms: tiotropium inhalation capsules

SUMMARY:
The objective of this study is to compare the bronchodilator efficacy and safety of tiotropium inhalation capsule (18 mcg once daily) and Atrovent MDI (2 puffs of 20 mcg q.i.d.) in patients with chronic obstructive pulmonary disease (COPD)

ELIGIBILITY:
Inclusion Criteria:

* COPD patients with an forced expiratory volume in one second (FEV1) <= 65% of predicted normal and FEV1 <= 70% of forced vital capacity (FVC)
* Male or female patients 40 years of age or older.
* Patient must have a smoking history of more than 10 pack-years. A pack-year is defined as the equivalent of smoking on pack of cigarettes per day for a year.
* Patient must be able to perform pulmonary function test as required in the protocol.
* Patient must be able to inhale medication from the handihaler device and should have a good technique of inhaling aerosol administered from MDI.
* All patients must sign an informed consent from prior to participation in the trail, prior to pre-study washout of their usual pulmonary medication.

Exclusion Criteria:

* Patient with significant disease other than COPD will be excluded. A significant disease is defined as a disease which in the opinion of the investigator may either put the patient at risk because of participation in the study or a disease which may influence the result of the study or the patient's ability to participate in the study.
* Patients with clinically significant abnormal baseline hematology, blood chemistry or urinalysis, if the abnormality defines a disease listed as an exclusion criterion will be excluded.
* All patients with a serum glutamic-oxaloacetic transaminase (SGOT) and serum glutamic-pyruvic transaminase (SGPT) twice the upper normal limit, bilirubin 150% or creatinine 125% of the upper normal limit will be excluded regardless of the clinical condition. Repeat laboratory evaluation will be not be conducted in these subjects.
* Patients with a recent history ( i.e. one year or less) of myocardial infarction.
* Patients with a recent history ( i.e. one year or less) of heart failure or patients with any cardiac arrhythmia requiring drug therapy.
* Patients with regular use of daytime oxygen therapy.
* Patients with known active tuberculosis.
* Patients with a history of cancer within the last five years. Patients with treated basal cell carcinoma are allowed.
* Patients with a history of life-threatening pulmonary, or history of cystic fibrosis or bronchiectasis.
* Patients who have undergone pulmonary resection or a thoracotomy for any reason.
* Patients with an upper respiratory tract infection in the past 2 weeks prior to the screening visit (= Visit 1) or during the baseline period of 2-weeks (run-in period).
* Patients with known hypersensitivity to anticholinergic drugs, lactose or any other component of the inhalation capsule delivery system.
* Patients with known symptomatic prostatic hypertrophy or bladder neck obstruction.
* Patients with known narrow-angle glaucoma.
* Patients who are being treated with cromolyn sodium or nedocromil sodium.
* Patients who are being treated with antihistamines.
* Patients using oral corticosteroid medication at unstable dosage (i.e. less than 6 weeks on a stable dose) or at a dose excess of the equivalent 10 mg of prednisone per day or 20 mg every day.
* Pregnant or nursing women or women of childbearing potential not using medically approved means of contraception (e.g. oral contraceptives, intrauterine devices, or diaphragm).
* Patients with a history of asthma, allergic rhinitis or atopy or who have a blood total eosinophil count >= 400 per microliter (males) or >= 320 per microliter (females). A repeat eosinophil count will not be conducted in these patients.
* Patients with a history and/or active alcohol or drug abuse.
* Patients who have taken an investigational drug on month or six half-lives (whichever is greater) prior to the screening visit (= Visit 1).

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2001-06; Primary Completion 2002-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline in trough forced expiratory volume in one second (FEV1) | baseline, day 29

SECONDARY OUTCOMES:
Change from baseline in forced expiratory volume in one second (FEV1), area under curve from 0 to 3 hours post drug administration | baseline, day 29
Change from baseline in forced vital capacity (FVC), area under curve from 0 to 3 hours post drug administration | baseline, day 29
Change from baseline in total score of patient evaluation questionnaire | baseline, day 29
Number of rescue medications | Up to day 29
Trough forced vital capacity (FVC) response | baseline, day 29
Number of patients with adverse events | up to day 29
Changes in vital signs (blood pressure, pulse rate) | up to day 29
Changes in electrocardiogram | up to day 29
Changes in safety laboratory tests | up to day 29